CLINICAL TRIAL: NCT03620929
Title: The Effect of Estrogen in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: Estrogen in the Prevention of Adhesion Reformation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yang Ling Ling, principal investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018FXHEC-KY025
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Asherman Syndrome
Keywords: estradiol
MeSH Terms: conditions — Gynatresia | interventions — Estradiol; Dydrogesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Having estrogen(Estradiol Valerate) after hysteroscopic adhesiolysis three months, all patients in this group will be treated with hormone therapy for 3 cycles; each cycle consists of estradiol 4mg per day for 21 days with addition of progestogen in the form of dydrogesterone 10mg per day for the last 7 days;
  Interventions: Drug: Estradiol Valerate
- Control group (No Intervention): Control group without estrogen treatment. A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.

INTERVENTIONS:
Drug: Estradiol Valerate — In all cases hormone therapy will be started from the day of operation, consisting of estradiol valerate at a dose of 4mg/d for 21 days, with the addition of dydrogesterone at a dose of 10 mg/d for the last 7 days of the estrogen therapy. After the withdrawal bleed, the hormone therapy will be repeated for another cycle. Second-look hysteroscopy will be carried out in the early proliferative phase, 4 weeks after the initial operation; a third-look hysteroscopy will be carried out 8 weeks after the initial operation. After assessment of the extent and severity of any reformed adhesion, hysteroscopic adhesiolysis will be carried out at the time of the second-look or third-look procedure, if adhesion had recurred.
  Other Names: dydrogesterone
  Arms: Experiment group

SUMMARY:
Asherman syndrome, which occurs after trauma to the basalis layer of the endometrium.It seems that the role of postoperative estrogen therapy in the prevention of recurrence of IU adhesions is still controversial. To investigate if estrogen therapy can prevent adhesion reformation after adhesiolysis.

After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: having estrogen after hysteroscopic adhesiolysis three months, all patients in this group will be treated with hormone therapy for 3 cycles; each cycle consists of estradiol 4mg per day for 21 days with addition of progestogen in the form of dydrogesterone 10mg per day for the last 7 days; and the control group without estrogen treatment. A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.

DETAILED DESCRIPTION:
Background information Asherman syndrome, which occurs after trauma to the basalis layer of the endometrium generally after endometrial curettage, may manifest as hypomenorrhea, amenorrhea, dysmenorrhea, infertility or recurrent miscarriage.

At present, hysteroscopic adhesiolysis is the recommended standard diagnostic method and treatment for IUA. Recurrence of uterine cavity adhesion post-operatively is frequently reported, especially in severe IUA patients. A number of strategies have been proposed to prevent recurrence of adhesion reformation, including the use of post-operative estrogen. However, it is still not known if estrogen therapy is indeed necessary or effective. In a prospective randomized study which evaluated the efficacy of estrogen in preventing IUA following hysteroscopic septal resection, it was found that estrogen did not have any benefit in reducing adhesion formation. In another RCT study on women with Asherman syndrome, there did not appear to be any difference in the recurrence of IUA and pregnancy rate between those who did or did not receive adjuvant hormonal medication. On the other hand, large doses of estrogen may result in endometrium fibrosis and inhibited endometrium receptivity.

It seems that the role of postoperative estrogen therapy in the prevention of recurrence of IU adhesions is still controversial. In this prospective, randomized, controlled study, we wish to determine if estrogen therapy is of benefit in preventing adhesion reformation after IUA for Asherman syndrome. As the effect may be different for subjects with different degrees of IUA, we propose to stratify the subjects into those with mild and severe IUAs.

Objectives To investigate if estrogen therapy can prevent adhesion reformation after adhesiolysis.

Patients The patients will be recruited from the hysteroscopy Center of the Fuxing Hospital, Beijing, China. Before the surgery all patients with suspected Asherman syndrome will undergo preoperative evaluations, including a detailed history of the menstrual pattern, any previous intrauterine surgery, reproductive history, as well as trans-vaginal ultrasonography. The severity and extent of intrauterine adhesions will be scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version). The inclusion criteria include [1] women aged 18-40 years; written consent obtained; and agreement to have second-look hysteroscopy. The exclusion criteria included:1 has received estrogen therapy within 3 month of enrolment. 2 suffers from leiomyoma, endometrial polyps, cancer, or polycystic ovarian syndrome (PCOS). 3.History of genital tuberculosis; and 4. contraindications for estrogen therapy.

Study Design After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: having estrogen after hysteroscopic adhesiolysis three months, all patients in this group will be treated with hormone therapy for 3 cycles; each cycle consists of estradiol 4mg per day for 21 days with addition of progestogen in the form of dydrogesterone 10mg per day for the last 7 days; and the control group without estrogen treatment. A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.

Power Calculation On the basis of the results of the two published retrospective cohort studies comparing the balloon and hormone therapy group (control group) in the prevention of adhesion reformation, in the mild intrauterine adhesion (AFS score 1~6), we estimate that the adhesion reformation rate the hormone therapy group is 10% and control group is 30%. Accepting a type 1 error (a) of 0.05, and a type 2 error (b) of 0.10, the number of subjects in each arm of the randomized, controlled trial would be 39. Assuming that the dropout rate is 20%, the total number of subject to be recruited would be 49 in each arm. In the severe intrauterine adhesion (AFS score7~12) group, we estimate that the adhesion reformation rate the hormone therapy group is 25% and control group is 50%. Accepting a type 1 error (a) of 0.05, and a type 2 error (b) of 0.10, the number of subjects in each arm of the randomized, controlled trial would be 37. Assuming that the dropout rate is 20%, the total number of subject to be recruited would be 44 in each arm.

Procedure Surgical procedure The surgery will be carried out by one of three experienced hysteroscopic surgeons with the use of a 4.5-mm rigid hysteroscope (Olympus) with 5% saline perfusion under 100 mm Hg pressure. The primary procedure will be performed under general anesthesia in a day surgery unit. Ultrasonographic guidance will be routinely used. Once the extent and severity of uterine adhesion has been assessed, the adhesions will be divided with the use of mono-polar instrument until normal uterine anatomy is achieved.

Postoperative treatments All subjects will be treated with oral antibiotic for 5 days. In all cases hormone therapy will be started from the day of operation, consisting of estradiol valerate at a dose of 4mg/d for 21 days, with the addition of dydrogesterone at a dose of 10 mg/d for the last 7 days of the estrogen therapy. After the withdrawal bleed, the hormone therapy will be repeated for another cycle. Second-look hysteroscopy will be carried out in the early proliferative phase, 4 weeks after the initial operation; a third-look hysteroscopy will be carried out 8 weeks after the initial operation. After assessment of the extent and severity of any reformed adhesion, hysteroscopic adhesiolysis will be carried out at the time of the second-look or third-look procedure, if adhesion had recurred. The surgeon who later performs the second-look and third-look hysteroscopy will be blinded to the randomization. All patients will be treated with hormone therapy for a total of three cycles.

ELIGIBILITY:
Inclusion Criteria:

patients with suspected Asherman syndrome

Exclusion Criteria:

* 1 has received estrogen therapy within 3 month of enrolment. 2 suffers from leiomyoma, endometrial polyps, cancer, or polycystic ovarian syndrome (PCOS). 3.History of genital tuberculosis; and 4. contraindications for estrogen therapy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
AFS score | 3 months
  The severity and extent of intrauterine adhesions will be scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version).

CONTACTS AND LOCATIONS:
Locations (1):
- Fuxing hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] March CM. Intrauterine adhesions. Obstet Gynecol Clin North Am. 1995 Sep;22(3):491-505. PMID 8524533
- [Background] ASHERMAN JG. Traumatic intra-uterine adhesions. J Obstet Gynaecol Br Emp. 1950 Dec;57(6):892-6. doi: 10.1111/j.1471-0528.1950.tb06053.x. No abstract available. PMID 14804168
- [Background] Schenker JG. Etiology of and therapeutic approach to synechia uteri. Eur J Obstet Gynecol Reprod Biol. 1996 Mar;65(1):109-13. doi: 10.1016/0028-2243(95)02315-j. PMID 8706941
- [Background] Schenker JG, Margalioth EJ. Intrauterine adhesions: an updated appraisal. Fertil Steril. 1982 May;37(5):593-610. doi: 10.1016/s0015-0282(16)46268-0. No abstract available. PMID 6281085
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Roy KK, Negi N, Subbaiah M, Kumar S, Sharma JB, Singh N. Effectiveness of estrogen in the prevention of intrauterine adhesions after hysteroscopic septal resection: a prospective, randomized study. J Obstet Gynaecol Res. 2014 Apr;40(4):1085-8. doi: 10.1111/jog.12297. Epub 2014 Feb 26. PMID 24612233
- [Background] Zhou Q, Wu X, Dai X, Yuan R, Qi H. The different dosages of estrogen affect endometrial fibrosis and receptivity, but not SDF-1/CXCR4 axis in the treatment of intrauterine adhesions. Gynecol Endocrinol. 2018 Jan;34(1):49-55. doi: 10.1080/09513590.2017.1328050. Epub 2017 May 20. PMID 28531361